CLINICAL TRIAL: NCT03386019
Title: The Efficacy of Lymphatic Massage on Lower Extremity Edema and Performance After Treadmill Exercise in Sprinter Compare to Static Stretching and Cold Water Immersion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201709058RINA
Record Dates: First submitted 2017-12-15; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-10

CONDITIONS: Post-exercise Lower Extremity Edema
Keywords: lymphatic massage; static stretching; cold water immersion
MeSH Terms: interventions — Manual Lymphatic Drainage; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: There will be a total of 4 different time points where outcome measures will be assessed including: baseline, immediately after pre-conditioning, immediately after treatment and 10 minutes after treatment. Once the participant completed the assessment of one treatment, another assessment session from one of the two remaining treatments will be scheduled in the following week, and the data collections for all three treatments will be finished in three consecutive weeks. This could ensure that all participants receive similar training schedules with similar training intensity within a fixed time period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sprinters (Experimental): Sprinters will be recruited from the track and field team of National Taiwan Normal University (NTNU) in this study. After individuals' enrollments and baseline data collections, all subjects will receive all three different treatments (massage, cold water immersion and static stretching) in randomized orders a week apart, respectively. Outcome measures are: visual analogue scale (VAS) score, lower leg volume, pressure pain threshold and horizontal jump distance. All measurements will be recorded at baseline, immediately after exercise, immediately after treatment, and 10 minutes after treatment as the follow up.
  Interventions: Other: Lymphatic massage; Other: Static stretching; Other: Cold water immersion

INTERVENTIONS:
Other: Lymphatic massage — One certified physical therapist will perform the massage regimens and techniques adapting from Swedish massage such as effleurage and petrissage that will be used in the massage group. Participants will first lay down in prone position, and the massage leg will be supported on the therapist's leg or on pillows with legs being positioned at approximately 30 degrees of knee flexion. This can promote venous return of the lower legs and also keep the ankle plantar flexors in a relative low muscle tension position. After positioning, long strokes will be applied from the distal to proximal part of gastrocnemius with approximately 20 repetitions and then 20 repetitions of circular strokes would be applied at the popliteal fossa. Finally, therapist will knead around participant's Achilles tendon for 10 repetitions.6 The combination of the techniques mentioned above will repeat 3 times in each subject, and the total duration of massage will be approximately 5 minutes.
Other: Static stretching — For the static stretching group, participants will perform the standing gastrocnemius stretches. First, participant stands facing a wall and put the stretched leg behind the body. Physical therapist will ask the participant to slightly flex the front leg, and keep back leg extended with heel on the ground. Both toes will be positioned pointing forward. Participant will then be asked to lunge forward slowly until the calf muscles on the back leg feeling stretched. Participant will hold in this position for 60 seconds and repeat 3 times.
Other: Cold water immersion — In the cold-water immersion group, participant's lower leg will be put in a bucket filled with cold water for 10 minute. The temperature of the water will be kept in 11-15 degrees Celsius.52 The water level should reach participant's fibular head to ensure complete immersion of the lower leg.

SUMMARY:
Background: Lower extremity edema is often seen after exercise in healthy individuals, especially sprinters, in sports physical therapy practice. Edema is defined as the excessive fluid accumulation in the interstitial space. Recent studies showed that there could be an increase in fluid up to 31.2 ml after a 15-minute running bout in healthy individuals. Fluid accumulation may be resulted from (1) high intensity training, (2) compression of blood and lymph vessels due to increased soft tissue tension and (3) the effect of gravity. Lower extremity edema not only causes great impact on athlete's recovery and performance, it could also lead to fibrosis, dysfunction and contracture. The pilot study showed that lower extremity edema not only existed post-exercise, and decreased ankle circumference was found after a 5-minute massage session, not only when compared to the status after exercise, but also when compared to the baseline (resting). The result also showed lower extremity edema may exist both during resting and after exercise. However, no studies to date investigated the solutions to decrease lower extremity edema during resting and after exercise in sprinters. Massage has been proven beneficial to athletes by increasing range of motion, promote recovery and increase skin blood flow, however, no study investigated the effect of massage on lower extremity edema and compared that to different common recovery modalities such as cold water immersion and static-stretching.

Purposes: To explore the effects of massage on sprinter's gastrocnemius after running on edema and strength with immediate and short-term follow ups.

Methods: This study will recruit both male and female sprinters age between 20-30 years old who participate in the event of 100, 200 and 400 meter sprints. After individuals' enrollments and baseline data collections, all subjects will receive all three different treatments (massage, cold water immersion and static stretching) in randomized orders a week apart, respectively. Outcome measures are: visual analogue scale (VAS) score, lower leg volume, pressure pain threshold and horizontal jump distance. All measurements will be recorded at baseline, immediately after exercise, immediately after treatment, and 10 minutes after treatment as the follow up. Descriptive statistics will be used for participants' characteristics. Three-way ANOVA (3 treatments x 4 times x 2 legs) with repeated measures design will be used to detect differences, and post-hoc analysis will be used when interactions are identified. p value of < .05 will be used in this study.

ELIGIBILITY:
Inclusion criteria:

1. 20-30 years-old of age.
2. Sprinters participate in 100-meter, 200-meter or 400-meter sprint events.
3. Trainings at least 5 days per week and at least 2 hours per day.

Exclusion criteria:

1. Lymphedema
2. Peripheral arterial disease
3. Chronic venous disease
4. Musculoskeletal injuries of the testing leg in recent 3 months (that would influence practice schedule)

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Lower leg volume | change from baseline to 10 minutes after treatment
  Lower leg volume was measured with water displacement method using volumeter. First, the volumeter was filled with water until it overflowed into the pitcher under the spout. Before each measurement, the pitcher was emptied, dried and placed back under the spout. The height of the chair was adjusted to ensure that the lower leg was completed immersed into water (the level of the water reached the mark). The pitcher filled with water collected from the volumeter was then weighed so that the volume of the lower leg could be quantified. Since the density of water was close to 1, the weight of the outflowed water was equal to the volume of the lower leg. To ensure that the assessor could measure the same site at all time periods, the same mark was used in each testing session.

SECONDARY OUTCOMES:
Pressure pain threshold | change from baseline to 10 minutes after treatment
  Pressure pain threshold was defined as the minimal amount of pressure that induced pain or discomfort. Participant was asked to lie in prone position with ankle sticking out of the edge of table to let the ankle slightly plantar flexed without resistance. The algometer was then placed at the muscle tendon junction of gastrocnemius on the testing leg. The assessor compressed the site with the algometer and gradually increasing pressure until the participant said "stop" whenever he or she started to feel pain or discomfort. At the same time, the second assessor read and recorded the value displayed on the algometer. Measurements were measured two times and the intervals between each measurement were around 5 seconds apart. These two readings were averaged and recorded for further data processing. The algometer showed good intra-rater reliability with an ICC of 0.96.
Perception of discomfort | change from baseline to 10 minutes after treatment
  Perception of discomfort such as tightness was assessed with visual analog scale (VAS), a grading scale range from 0 to 100 mm. 0 mm represented no pain or discomfort at all and 100 mm represented the greatest amount of pain or discomfort imaginable. Participant drew a line that intersects the grading scale to show the amount of pain or discomfort that he or she experienced at that moment. The assessor then used a ruler to measure the length from 0 mm to the intersecting line and recorded the value. Perception of discomfort was assessed at each time point.
Horizontal jump distance | change from baseline to 10 minutes after treatment
  Horizontal jump or standing long jump was a common performance test to examine the athlete's power and aerobic capacity. The athlete started from a standing position and were then asked to jump forward as far as they could by bending their knees and swinging both arms. A starting line was drawn and the expected landing region was placed with mat to prevent any possible injuries occurred. After the jump, the distance from starting line to where the participant's heel landed was measured. If the participant's heels were landed unleveled, the heel that was closer to the starting line was measured. The participant jumped twice in each time point. The jump distances in the same time point was then averaged.

CONTACTS AND LOCATIONS:
Locations (1):
- School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No